CLINICAL TRIAL: NCT02356224
Title: Pharmacokinetics, Pharmacodynamics, Safety and Tolerability Study Following Single Dose of SHR3824 in Healthy Subjects
Brief Title: The PK/PD Study of Single Dose of SHR3824 in Healthy Volunteers
Acronym: SHR3824
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR3824-101
Record Dates: First submitted 2015-01-29; First posted 2015-02-05 (Estimated); Last update posted 2015-02-05 (Estimated); Status verified 2014-12

CONDITIONS: Type 2 Diabetes
Keywords: SHR3824 Type 2 diabetes mellitus SGLT2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — henagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (7):
- Cohort 1 (Experimental): SHR3824 2.5 mg/day or placebo.
  Interventions: Drug: SHR3824; Drug: Placebo
- Cohort 2 (Experimental): SHR3824 5 mg/day or placebo. The actual dose (mg) level selected for each cohort may be modified based on evaluation of preliminary safety, pharmacokinetic and pharmacodynamic data from previous cohorts.
  Interventions: Drug: SHR3824; Drug: Placebo
- Cohort 3 (Experimental): SHR3824 10 mg/day or placebo. The actual dose (mg) level selected for each cohort may be modified based on evaluation of preliminary safety, pharmacokinetic and pharmacodynamic data from previous cohorts.
  Interventions: Drug: SHR3824; Drug: Placebo
- Cohort 4 (Experimental): SHR3824 25 mg/day or placebo. The actual dose (mg) level selected for each cohort may be modified based on evaluation of preliminary safety, pharmacokinetic and pharmacodynamic data from previous cohorts.
  Interventions: Drug: SHR3824; Drug: Placebo
- Cohort 5 (Experimental): SHR3824 50 mg/day or placebo. The actual dose (mg) level selected for each cohort may be modified based on evaluation of preliminary safety, pharmacokinetic and pharmacodynamic data from previous cohorts.
  Interventions: Drug: SHR3824; Drug: Placebo
- Cohort 6 (Experimental): SHR3824 100 mg/day or placebo. The actual dose (mg) level selected for each cohort may be modified based on evaluation of preliminary safety, pharmacokinetic and pharmacodynamic data from previous cohorts.
  Interventions: Drug: SHR3824; Drug: Placebo
- Cohort 7 (Experimental): SHR3824 200 mg/day or placebo. The actual dose (mg) level selected for each cohort may be modified based on evaluation of preliminary safety, pharmacokinetic and pharmacodynamic data from previous cohorts.
  Interventions: Drug: SHR3824; Drug: Placebo

INTERVENTIONS:
Drug: SHR3824 — A tablet of 2.5 mg, 5 mg, 10 mg, 25 mg, 50mg, 100mg, 200 of SHR3824 taken for single dose.
  Other Names: Henagliflozin
Drug: Placebo — A tablet of 2.5 mg, 5 mg, 10 mg, 25 mg, 50mg, 100mg, 200 of Placebo taken for single dose.

SUMMARY:
SHR3824 is a novel inhibitor of renal sodium-glucose cotransporter 2, allows an insulin-independent approach to improve type 2 diabetes hyperglycemia. In this single-dose study the investigators evaluated the safety, tolerablity and PK/PD profiles of SHR3824 in healthy subjects.

ELIGIBILITY:
Inclusion criteria:

* Chinese male and female subjects aged 18 to 45 years.
* BMI:18 -25 kg/m2 .
* Healthy according to medical history, physical examination findings, 12-lead ECG findings, and clinical laboratory evaluations.

Exclusion criteria:

* History of or current clinically significant medical illness as determined by the Investigator.
* History of clinically significant allergies, especially known hypersensitivity or intolerance to lactose.
* Pregnancy or breastfeeding .
* Significant acute or chronic medical illness, including renal impairment, or recent surgery.
* Donation of blood or plasma within the 4 weeks prior to the start of the study or acception of blood transfusion within 8 weeks.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2013-06; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Total 24-hour urinary glucose excretion as a measure of pharmacodynamic effect. | 24h after dosing
SHR3824 and its metabolites of concentrations to characterize SHR3824 harmacokinetics. | Up to 72h after dosing

SECONDARY OUTCOMES:
The number of patients with adverse events as a measure of safety and tolerability | up to day 72h after dosing

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Xuhui Central Hospital, Shanghai, Shanghai Municipality, China